CLINICAL TRIAL: NCT06125769
Title: LIver TrAnspLantation for Non-resectable Peri-HIlar cholangioCArcinoma (LITALHICA)
Acronym: LITALHICA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Sanitaria Ospedaliera (Other)
Collaborators: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Principal Investigator, Enrico Gringeri, Associate Professor, Azienda Sanitaria Ospedaliera
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOP 3007
Record Dates: First submitted 2023-10-30; First posted 2023-11-09 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Perihilar Cholangiocarcinoma
Keywords: Liver transplantation
MeSH Terms: conditions — Klatskin Tumor | interventions — Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study population (Experimental): Candidates will be evaluated by the Multidisciplinary Group after routine radiological studies (CT, MRI, PET-MRI/CT).
  Patients will receive 6 months of standard of care chemotherapy and undergo PET-MRI with FDG to exclude the presence of extrahepatic disease.
  Following completion of therapy, patients will undergo radiological restaging. If the disease is resectable, the patient will be considered for curative-intent surgical resection; if not, the patients will be evaluated by the Center's Multidisciplinary Transplantation Group. Patients will continue chemotherapy until a compatible liver becomes available. If there are no further contraindications, exploratory laparotomy and surgical nodal staging of the tumor will be performed at the time of transplantation. If there are no signs of extrahepatic disease, transplantation will be conducted according to institutional protocols.
  Interventions: Procedure: Liver transplantation

INTERVENTIONS:
Procedure: Liver transplantation — Patients will undergo liver transplantation according to the standard procedures of the institutional Center's protocol (cadaveric or living donor transplantation, whole or partial liver). Liver transplantation is preceded by an exploratory laparotomy with clinical evaluation and frozen section examination of lymph nodes in the hepatoduodenal ligament and along the common hepatic artery/celiac axis.

SUMMARY:
LITALHICA is a prospective non-randomized study aimed at exploring the outcome of liver transplantation in selected patients with unresectable perihilar cholangiocarcinoma (pCCA) after treatment with standard of care chemotherapy, in terms of overall survival and quality of life. Additionally, the study aims to identify pre-transplant biological markers and clinical factors that can stratify patients with the best post-transplant prognosis. Finally, the study aims to investigate the role of preoperative PET-MRI, especially in relation to lymph node locations, by correlating the results with histological examination after hilar lymphadenectomy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pCCA (transcatheter biopsy or brush cytology, CA 19-9 > 100 mg/mL and/or a mass on cross-sectional imaging with a malignant appearing stricture on cholangiography, or biliary ploidy with a malignant appearing stricture on cholangiography)
* Disease considered unsuitable for hepatic resection based on tumor location and extent or underlying liver dysfunction
* Absence of major vascular invasion, extrahepatic disease, or involvement of regional lymph nodes detected on radiological study
* No evidence of extrahepatic metastatic disease after chest-abdomen-pelvis CT and PET-MR (or PET-CT)
* Unresectable tumor above cystic duct (pancreatoduodenectomy for microscopic involvement of CBD) or resectable pCCA arising in PSC
* Radial tumor diameter <3 cm
* At least six months have passed since the first diagnosis of pCCA to the date of inclusion on the liver transplant waiting list
* The patient has received at least six months of standard of care (SOC) chemotherapy, achieving disease stability or partial response (according to RECIST criteria version 1.1) at the time of listing for transplantation
* Absence of medical or surgical contraindication to liver transplantation
* Signed informed consent, and expected patient cooperation for treatment and follow-up, must be obtained and documented according to good clinical practice and national/local regulations

Exclusion Criteria:

* Diagnosis of intrahepatic cholangiocarcinoma (iCCA)
* Uncontrollable infection
* Prior radiotherapy or chemotherapy
* Prior biliary surgical resection or attempted surgical resection
* Diameter of tumor >3cm
* Presence of intra-hepatic metastases
* Present or past evidence of extrahepatic metastatic disease
* Transperitoneal biopsy (including percutaneous ecography-guided FNA)
* Prior neoplasms, except those treated curatively for more than 5 years without recurrence
* Substance abuse and medical, psychological, or social conditions that may interfere with the patient's participation in the study or with the evaluation of study outcomes
* Pregnant or breastfeeding women
* Medical-surgical contraindications for liver transplantation
* Any reason for which, in the investigator's judgment, the patient should not participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2033-11-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 3 and 5 years
  Survival from time of transplantation to time of death or last follow up

SECONDARY OUTCOMES:
Overall survival comparison with chemotherapy alone | 3 years
  Comparison of 3-year survival between patients enrolled in the LITALHICA study and survival of a population balanced for prognostic factors and disease characteristics from the database of the Veneto Oncological Institute (IOV)
Progression-Free Survival (PFS) | 3 and 5 years
  Survival from time of transplantation to time of death or first evidence of progression of disease
Overall survival from the time of recurrence | 5 years
  Survival from time of recurrence to time of death or last follow up
Progression-free survival comparison with chemotherapy alone | 3 years
  Comparison of 3-year progression-free survival between patients enrolled in the LITALHICA study and progression-free survival of a population balanced for prognostic factors and disease characteristics from the database of the Veneto Oncological Institute (IOV)
Biological markers | 5 years
  Correlation of overall survival and recurrence with tissue and circulating biological markers (immunohistochemistry, proteomics, circulating tumor cells, circulating tumor DNA, new molecular markers)
Morbidity | 90 days
  Morbidity at 90 days (according to Clavien-Dindo and Comprehensive Complication Index, CCI)
Cancer-related mortality | 3 and 5 years
  Risk of mortality with sole relation to death by tumor progression
Drop out | 5 years
  Percentage of patients who do not complete the procedure (drop-out) stratified by cause
Concordance of surgical and PET/MRI staging | Perioperative
  Asses if lymph nodes described as suspicious at the preoperative PET-MRI confirm to be pathological at the histological evaluation after lymphadenectomy of the hepatic hilum and exploratory laparotomy
Quality of life assessed using EORTC QLQ-C30 | 5 years
  Quality of life assessed using EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer QLQ Core Questionnaire) 30 items questionnaire (scale 1-4 or 1-7, 1 being the lowest and 4 or 7 the highest, accordingly)
Quality of life assessed using FACT-Hep questionnaire | 5 years
  Quality of life assessed using FACT-Hep questionnaire (Functional Assessment of Cancer Therapy - Hepatobiliary) questionnaire about quality of life in the last 7 days (scale 0-4, 0 being the lowest and 4 the highest)

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Gringeri, Prof., Principal Investigator — Azienda Ospedale Università di Padova
Locations (1):
- Azienda Ospedale Università di Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No